CLINICAL TRIAL: NCT02358720
Title: Single-fraction IMRT Versus External Beam Radiotherapy for Patients With Spine Bone Metastases
Acronym: SMART
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART
Record Dates: First submitted 2015-01-27; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Pain
Keywords: bone metastases
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: single fraction IMRT with 1 x 24 Gy (Experimental): single fraction IMRT with 1 x 24 Gy on bone metastasis
  Interventions: Radiation: Arm A
- B: fractionated RT with 10 x 3 Gy (Active Comparator): fractionated RT with 10 x 3 Gy on bone metastasis
  Interventions: Radiation: Arm B

INTERVENTIONS:
Radiation: Arm A — 1x24Gy high dose IMRT on spinal bone metastasis
  Arms: A: single fraction IMRT with 1 x 24 Gy
Radiation: Arm B — fractionated conformal RT 10 x 3 Gy on spinal bone metastasis
  Arms: B: fractionated RT with 10 x 3 Gy

SUMMARY:
This study is a prospective, randomized, monocentre, controlled explorative study in the parallel-group design to determine the pain relief after RT of patients with spinal bone metastases. Thereby two different techniques were evaluated: single fraction IMRT with 1 x 24 Gy versus fractionated RT with 10 x 3 Gy. Prior to their enrolment into the study, the patients will undergo a staging of the vertebral column in connection with their radiation-planning computed tomography (CT) and MRI to measure the myelon dimension. After the baseline results have been recorded, the patients will be randomized into one of the two groups: single-fraction IMRT 1 x 24 Gy (n = 30) or fractionated RT 10 x 3 Gy (n = 30). The target parameters will be measured and recorded at baseline, at the end of RT (t1) and twelve weeks (t2) and six months following the end of the irradiation period (t3).

DETAILED DESCRIPTION:
The patients will be given information on the study by the medical personnel of the Radiotherapy Department in connection with the planning of the RT schedule (approximately 1-2 weeks prior to the start of RT). If they are interested in participating in the study, the potential study candidates will be given the Patient Information sheet including the Declaration of Informed Consent, with the request that they reread the information carefully and if they consent to the conditions return the signed declaration when they attend the next appointment. The patients will be given the opportunity to ask the study staff further questions. Among the preconditions for participation in the study is the condition that no metastatic spinal cord compression (tumor distance > 3 mm to myelon) of the metastasized vertebral body is detected in MRI recorded in the course of planning procedure. A block randomization procedure shall be used to ensure the even distribution of the patients into the two intervention groups, stratified to baseline pain level. The patients shall then be assigned 1:1 to one of the two treatment groups on the basis of the baseline measurements. The randomization procedure shall be carried out by a central office. The study personnel responsible for the recruitment and baseline measurements shall have no access to the randomization list, and the study director no influence on the recruitment of the patients. The recruitment phase shall be concluded with the attainment of the planned number of patients (60 patients in total). It shall last twelve months, and is scheduled to start in December 2014. Regular study participation shall end six months after enrolment into the study or, where applicable, with the respective patient's death. The aim of the trial was to evaluate the pain relief after RT of patients with spinal bone metastases. Thereby two different techniques were evaluated: single fraction IMRT with 1 x 24 Gy versus fractionated RT with 10 x 3 Gy. The primary endpoint was defined as pain relief > 2 points according to visual analog scale (VAS) measured at the irradiated region up to three months after the end of RT (t2). Secondary endpoints were quality of life (QoL), fatigue, pain, overall survival, bone survival, local control, pathological fracture, and neurological deficit. The baseline examination shall be carried out on the first day of radiotherapy prior to the start of therapy and is scheduled to comprise the comprehensive recording of the sociodemographic data, the recording of the current pain situation, the fear of suffering fractures, the quality of life, and the current degree of fatigue. The follow-up examinations shall take place after the end of radiotherapy (day of the last fraction) and twelve weeks and six months after radiotherapy, measuring those parameters recorded at the baseline examination. The further follow-up examinations shall correspond to those carried out as standard after-care investigations.

The secondary endpoints such as fatigue, quality of life, and anxiety shall be recorded using validated questionnaires (EORTC QLQ FA13 (11), EORTC QLQ BM22 (12) and the questionnaire to record stress in cancer patients (FBK) according to Book et al. (13). All patients will also be asked to record their pain history using a pain diary (documentation of medication daily during treatment, once weekly after the end of treatment, VAS pain scale). Furthermore, the local control was assessed by means of CT images taken prior to, three and six months after RT. The pain response was documented on the VAS (range 0-10). Complete response (CR) was defined as VAS = 0 after three and six months, partial response (PR) as an improvement by at least two score points after three and six months, according to the international consensus response categories by Chow et al. (14). Overall survival (OS) was defined as time from initial diagnosis until death, bone survival as time from initial diagnosis of spinal bone metastasis until death.

Radiotherapy Immobilization was assessed with Aquaplast head mask®, vacuum mattress and Wingstep®. On the basis of the planning-CT risk organs and clinical target volume (CTV) were contoured. CTV confirmed planning target volume (PTV). The dose of PTV occured at the 80%-isodose, encircling the PTV. The RT procedure in group A was conducted as IMRT (Tomotherapy or Step-and-shoot IMRT) 24 Gy in a single-fraction occured at the 80%-isodose. In group B, RT was performed as irradiation of the involved vertebral body as well as the ones immediately above and below to a total-dose of 30 Gy with a single daily dose of 3 Gy using 6 MV individually-formed beams (Linac, multileaf collimator) after CT-scan based 3D planning. The tolerance doses of organs at risk were used according RTOG 0631 study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed tumor diagnosis, with secondary diagnosed solitary/multiple spinal bone metastases
* Indication for RT of the spinal bone metastases
* Maximal two irradiated vertebral-bodies per region
* Maximal two different vertebral regions
* Age: between 18 and 80 years
* Karnofsky index (10) ≥ 70
* Signed Declaration of Informed Consent
* Tumor distance > 3 mm to myelon

Exclusion Criteria:

* Multiple myeloma or lymphoma
* Significant neurological or psychiatric disorders, including dementia and epileptic seizures
* Earlier RT at the current irradiated site
* Other severe disorders that in the judgement of the study director may prevent the patient's participation in the study
* Lacking or diminished legal capacity
* Any medical of psychological condition that the study director considers a preventive factor for the patient's ability to complete the study or to adequately
* understand the scope of the study and to give his/her consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
pain relief, as measured by visual analog scale (VAS) | 3 months after therapy completed
  The primary endpoint was defined as pain relief > 2 points according to visual analog scale (VAS) measured at the irradiated region up to three months after the end of RT

SECONDARY OUTCOMES:
quality of life measured on an EORTC BM22 questionnaire | 3 and 6 months after therapy completed
  Secondary endpoints were quality of life (QoL) measured on an EORTC BM22 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Harald Rief, MD, PhD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- Dept of Radiation Oncology, University of Heidelberg, Germany, Heidelberg, Germany, Germany

REFERENCES:
- [Background] Coleman RE. Metastatic bone disease: clinical features, pathophysiology and treatment strategies. Cancer Treat Rev. 2001 Jun;27(3):165-76. doi: 10.1053/ctrv.2000.0210. PMID 11417967
- [Background] Chung Y, Yoon HI, Kim JH, Nam KC, Koom WS. Is helical tomotherapy accurate and safe enough for spine stereotactic body radiotherapy? J Cancer Res Clin Oncol. 2013 Feb;139(2):243-8. doi: 10.1007/s00432-012-1321-0. Epub 2012 Oct 2. PMID 23052695
- [Background] Nguyen QN, Shiu AS, Rhines LD, Wang H, Allen PK, Wang XS, Chang EL. Management of spinal metastases from renal cell carcinoma using stereotactic body radiotherapy. Int J Radiat Oncol Biol Phys. 2010 Mar 15;76(4):1185-92. doi: 10.1016/j.ijrobp.2009.03.062. Epub 2009 Jul 23. PMID 19632064
- [Background] Ryu S, Pugh SL, Gerszten PC, Yin FF, Timmerman RD, Hitchcock YJ, Movsas B, Kanner AA, Berk LB, Followill DS, Kachnic LA. RTOG 0631 phase 2/3 study of image guided stereotactic radiosurgery for localized (1-3) spine metastases: phase 2 results. Pract Radiat Oncol. 2014 Mar-Apr;4(2):76-81. doi: 10.1016/j.prro.2013.05.001. Epub 2013 Jun 4. PMID 24890347
- [Background] Janjan N, Lutz ST, Bedwinek JM, Hartsell WF, Ng A, Pieters RS Jr, Ratanatharathorn V, Silberstein EB, Taub RJ, Yasko AW, Rettenmaier A; American College of Radiology. Therapeutic guidelines for the treatment of bone metastasis: a report from the American College of Radiology Appropriateness Criteria Expert Panel on Radiation Oncology. J Palliat Med. 2009 May;12(5):417-26. doi: 10.1089/jpm.2009.9633. PMID 19416037
- [Derived] Sprave T, Verma V, Forster R, Schlampp I, Hees K, Bruckner T, Bostel T, El Shafie RA, Welzel T, Nicolay NH, Debus J, Rief H. Local response and pathologic fractures following stereotactic body radiotherapy versus three-dimensional conformal radiotherapy for spinal metastases - a randomized controlled trial. BMC Cancer. 2018 Aug 31;18(1):859. doi: 10.1186/s12885-018-4777-8. PMID 30170568
- [Derived] Sprave T, Verma V, Forster R, Schlampp I, Bruckner T, Bostel T, Welte SE, Tonndorf-Martini E, Nicolay NH, Debus J, Rief H. Randomized phase II trial evaluating pain response in patients with spinal metastases following stereotactic body radiotherapy versus three-dimensional conformal radiotherapy. Radiother Oncol. 2018 Aug;128(2):274-282. doi: 10.1016/j.radonc.2018.04.030. Epub 2018 May 26. PMID 29843899
- [Derived] Rief H, Katayama S, Bruckner T, Rieken S, Bostel T, Forster R, Schlampp I, Wolf R, Debus J, Sterzing F. High-dose single-fraction IMRT versus fractionated external beam radiotherapy for patients with spinal bone metastases: study protocol for a randomized controlled trial. Trials. 2015 Jun 9;16:264. doi: 10.1186/s13063-015-0761-7. PMID 26054533